CLINICAL TRIAL: NCT02751268
Title: Effect of Infraorbital and Infratrochlear Nerve Block on Emergence Agitation in Patients Undergoing Septorhinoplasty: A Randomized Controlled Trial
Brief Title: Effect of Infraorbital and Infratrochlear Nerve Block on Emergence Agitation in Patients Undergoing Septorhinoplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Armed Forces Hampyeong Hospital (Other)
Responsible Party: Principal Investigator, Hoon Choi, M.D. Department of Anesthesiology and Pain Medicine, Armed Forces Hampyeong Hospital, Armed Forces Hampyeong Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AFMC-16028-IRB-16-021
Record Dates: First submitted 2016-04-24; First posted 2016-04-26 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Emergence Agitation; Pain
Keywords: infraorbital nerve block; infratrochlear nerve block; septorhinoplasty; general anesthesia; postoperative analgesia
MeSH Terms: conditions — Emergence Delirium; Pain | interventions — Saline Solution; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): placebo for the realization of infraorbital and infratrochlear block
  Interventions: Drug: Normal Saline
- Ropivacaine (Active Comparator): ropivacaine for the realization of infraorbital and infratrochlear block
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Normal Saline — Bilateral infraorbital and infratrochlear nerve block before general anesthesia with normal saline
  Arms: Control
Drug: Ropivacaine — Bilateral infraorbital and infratrochlear nerve block before general anesthesia with 0.5% ropivacaine
  Arms: Ropivacaine

SUMMARY:
The purpose of this study is to determine whether bilateral infraorbital and infratrochlear nerve block in patients undergoing septorhinoplasty are effective in preventing emergence agitation.

DETAILED DESCRIPTION:
Emergence agitation is a postanesthetic phenomenon characterized as confusion, disorientation and violent behavior. Although its etiology is not well understood, risk factors associated with the condition include pain and ENT (ear, nose and throat) surgery. Bilateral infraorbital and infratrochlear nerve block in patients undergoing septorhinoplasty is effective in treating postoperative pain. The investigators have designed this study to evaluate the effect of infraorbital and infratrochlear nerve block on emergence agitation in patients undergoing septorhinoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Septorhinoplasty
* American Society of Anesthesiologists (ASA) classification I-II
* Written informed consent

Exclusion Criteria:

* ASA classification greater than III
* Allergy to ropivacaine
* Incapability to give consent
* Chronic pain
* Coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Emergence agitation | 2 hours after surgery
  Emergence agitation is measured by Riker Sedation-Agitated Scale (RASS) and is defined as RASS=5-7

SECONDARY OUTCOMES:
Pain intensity | 2, 8, 24, 48 hours after surgery
  0-10 numerical rating scale (NRS) : from 0 = no pain to 10 = worst pain imaginable
Patient satisfaction | 48 hours after surgery
  1-5 scale (1: very unsatisfactory, 2: rather unsatisfactory, 3: fair, 4: rather satisfactory, 5: very satisfactory)

CONTACTS AND LOCATIONS:
Overall Officials: Hoon Choi, M.D., Principal Investigator — Armed Forces Hampyeong Hostpital
Locations (1):
- Armed Forces Hampyeong Hospital, Geumgyeri, Haebo-myeon, Hampyeong-gun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HJ, Kim DK, Kim HY, Kim JK, Choi SW. Risk factors of emergence agitation in adults undergoing general anesthesia for nasal surgery. Clin Exp Otorhinolaryngol. 2015 Mar;8(1):46-51. doi: 10.3342/ceo.2015.8.1.46. Epub 2015 Feb 3. PMID 25729495
- [Background] Boselli E, Bouvet L, Augris-Mathieu C, Begou G, Diot-Junique N, Rahali N, Vertu-Ciolino D, Gerard C, Pivot C, Disant F, Allaouchiche B. Infraorbital and infratrochlear nerve blocks combined with general anaesthesia for outpatient rhinoseptoplasty: A prospective randomised, double-blind, placebo-controlled study. Anaesth Crit Care Pain Med. 2016 Feb;35(1):31-36. doi: 10.1016/j.accpm.2015.09.002. Epub 2015 Nov 5. PMID 26549134